CLINICAL TRIAL: NCT05226754
Title: Study Design of the Diacerein Effect on Inflammatory Response in Patients With Covid-19: a Randomized, Placebo-controlled, Double-blind Trial.
Brief Title: Study Design of the Diacerein in Patients With Covid-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, Director, Brazilian Heart Study Group, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50440921.6.0000.5404
Record Dates: First submitted 2022-02-02; First posted 2022-02-07 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: COVID-19; Diacerein; Inflammatory Cytokine; Clinical Trial
MeSH Terms: conditions — COVID-19 | interventions — diacerein; Lactose; stearic acid

STUDY DESIGN:
Intervention Model Description: After enrolment, patients will be randomized (n=20 per group) 1:1 to receive either diacerein 50 mg or placebo treatment every 12 hours for 10 days. The research electronic data capture (REDCap) platform will be used as a randomization system. Patients, investigators and other support staff will be blinded to the experimental therapy. The study drug, diacerein (Artrodar®-capsules 50mg) and placebo capsules (lactose and magnesium stearate), will be similar in size and appearance to maintain blinding. All laboratory analyses will be performed blinded to the treatment. Identification of the study drug will only occur after locking the dataset.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Active Comparator): diacerein 50 mg (capsules) every 12 hours for 10 days
  Interventions: Drug: Diacerein
- GROUP B (Placebo Comparator): placebo capsules (lactose and magnesium stearate)
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: Diacerein — After enrolment, patients will be randomized (n=20 group A) to receive diacerein capsules 50 mg every 12 hours for 10 days.
  Other Names: Artrodar®-capsules 50mg
  Arms: GROUP A
Drug: placebo capsules — After enrolment, patients will be randomized (n=20 group A) to receive placebo capsules (lactose and magnesium stearate) every 12 hours for 10 days.
  Other Names: lactose and magnesium stearate
  Arms: GROUP B

SUMMARY:
This is a randomized, placebo-controlled, double-blind trial pilot study. This study will include individuals over 18 years of age who have been hospitalized with a confirmed diagnosis of COVID-19 to assess whether DIACEREIN treatment is safe and effective in controlling or decreasing inflammation in the body and viral load (amount of virus in the body in these patients).

DETAILED DESCRIPTION:
Study Design This is a randomized, placebo-controlled, double-blind trial pilot study designed to verify whether diacerein attenuates systemic inflammatory response in hospitalized patients with COVID-19. This study has been reviewed and approved by the Ethics Committee of the State University of Campinas (CAAE: 50440921.6.0000.5404).

Study Population Forty patients with a confirmed diagnosis of COVID-19 will be enrolled in the study. The patients will be identified as those admitted to either Hospital Estadual Sumaré (Sumaré, Brazil) and Unicamp Clinical Hospital (Campinas, Brazil). After enrolment, patients will be randomized (n=20 per group) in a 1:1 fashion to receive either diacerein 50mg or placebo treatment every 12 hours for 10 days.

Recruitment All patients admitted with COVID-19 who meet the inclusion and exclusion criteria will be invited to participate in the study. After reading and signing the informed consent form, the patient will be randomly allocated to two treatment arms.

Randomization and Blinding After enrolment, patients will be randomized (n=20 per group) 1:1 to receive either diacerein 50 mg or placebo treatment every 12 hours for 10 days. The research electronic data capture (REDCap) platform will be used as a randomization system. Patients, investigators and other support staff will be blinded to the experimental therapy. The study drug, diacerein (Artrodar®-capsules 50mg) and placebo capsules (lactose and magnesium stearate), will be similar in size and appearance to maintain blinding. All laboratory analyses will be performed blinded to the treatment. Identification of the study drug will only occur after locking the dataset.

Trial Intervention After randomization, patients allocated to the active treatment will receive 1 capsule of diacerein (Artrodar®, 50mg) orally every 12 hours for 10 days. Patients randomized to the placebo group will receive 1 capsule (lactose and magnesium stearate) orally every 12 hours for 10 days. There will be a dose adjustment of study medication (diacerein or placebo) to 1 capsule every 24 hours (decreased diacerein to 50 mg every 24 hours instead of every 12 hours) in participants who experience acute kidney injury with a rate of estimated glomerular filtration rate <30mL/min or requiring renal replacement therapy. If renal replacement therapy is required, the study drug will be administered immediately after dialysis.

If the patient is intubated, the diacerein or placebo capsules will be opened and their contents will be placed in previously cleaned and properly identified nylon sachets. The sachet content will be dissolved in 10 to 20ml of distilled water in a 20ml syringe at the time of administration by the nursing in the presence of a researcher. The trial intervention will not delay or affect the patient's clinical management in accordance with local centre policies.

Laboratory analyses On admission, the first blood sample will be collected before the first dose of study drug (Day 0), and then three and ten hours after the drug administration. Blood samples will also be collected on the second (Day 2), fifth (Day 5) and tenth (Day 10) day of treatment. With the exception of samples obtained on admission, blood samples will be collected after a 12-hour fast. Immediately after collection, all samples will be centrifuged at 3,500 rpm and frozen in liquid nitrogen for single batch processing. Inflammatory cytokines (c-reactive protein, IL-1β, IL-6, IL-8, IL-10, IL-12p70, IFN-α2, IFN-β, IFN-γ, TNF-α, IP-10 GM-CSF) will be measured by multiplex immunoassay (Bio-Plex 200®, Bio-Rad) as well other markers such as troponin-T and D-dimer measurements.

Study Endpoints The endpoints are the change in the serum levels of cytokines, troponin-T and D-dimer from Day 0 to Day 5 of hospitalization, and from Day 0 to Day 10, as well as the area under the curve considering all measurements from Day 0 to Day 10.

Secondary endpoints include (i) time to clinical deterioration defined as time from randomization to mortality or worsening of the World Health Organization (WHO) Clinical Progression Scale, assessed by the increase of two points in this scale; (ii) cumulative incidence of adverse events; (iii) cumulative incidence of severe adverse events.

Diacerein Bioavailability The bioavailability of diacerein and its active metabolite, rhein, will be evaluated in the serum of patients randomized to diacerein treatment in order to assure the bioavailability in COVID-19 patients. It will be used samples from Day 0 and timepoints: soon before, three and ten hours after the study drug administration. All patients will have these samples collected to maintain study blinding. Serum diacerein and rhein concentrations will be determined by liquid chromatography-tandem mass spectrometry at the end of the study.

Sample Size Calculation As there are no data available on the effect of diacerein on the inflammatory response in patients with COVID-19 the sample size was empirically established at 40 subjects in a conservative expectation of small standardized effect size (0.2). Therefore, we decided to carry out a pilot sample with 40 patients (n=20 per arm of the study) with outcomes from systemic inflammatory response and safety.

The Safety Analysis Population Applied to all randomized patients who received at least one dose of diacerein. The safety assessment will be based on the cumulative incidence of safety outcomes, adverse events, physical examinations, vital signs, and safety laboratory tests. The primary safety endpoint will be the time between randomization and the first occurrence.

Statistical Analysis Continuous variables will be represented by the median and the associated interquartile range. Categorical variables will be presented as absolute frequency (n) and relative frequency (%). Summary statistical data (mean, standard deviation, median, minimum and maximum) will be provided by the treatment group for demographic and baseline characteristics using a chi-square test (e.g., categorical variables) and one-way analysis of variance (ANOVA) model with treatment as a factor (e.g., continuous variables). In addition, demographics and baseline characteristics will be compared across treatment groups for the intention to treat (ITT) population. The significance of this test will be used as an initial assessment for the satisfaction of randomization.

Concentrations of plasma pro-inflammatory cytokines will be considered as efficacy endpoints. The groups will be compared by the changes in admission (Day 0) versus assessment days (Day 2, Day 5 and Day 10). Also, comparison between the areas under the curve for each of the parameters from Day 0 to Day 10. Continuous variables with normal and non-parametric distribution will be compared by analysis of covariance (ANCOVA) or by analysis of rank of variance (RANKOVA) adjusted by baseline values to mitigate the regression toward the mean.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either sex (≥18 years of age) with a diagnosis of COVID-19 infection, confirmed by positive polymerase chain reaction PCR reaction.
* Patient or his/her legal representative provide written informed consent prior to the start of the study.

Exclusion Criteria:

* Patients already hospitalized and on mechanical ventilation for over 48 hours;
* Pregnant or breastfeeding women;
* Contraindication for the use of diacerein or history of diacerein hypersensitivity;
* End-stage renal disease requiring renal replacement therapy;
* Chronic liver disease and/or ALT and AST ≥5 times the normal upper reference limit;
* Any active underlying malignancy;
* Currently enrolled in another research study;
* Peripheral capillary oxygen saturation/fraction of inspired oxygen ratio <100;
* Use of high dose of >1.0 mcg/kg/min of norepinephrine or need for rescue therapy with vasopressin;
* Bacterial or fungal infection, except for mild cutaneous infection or sinus infection.
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if they were to participate in the study;
* Clinically relevant serious co-morbid medical conditions including, but not limited to, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, severe hepatic impairment, active central nervous system (CNS) disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV), active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements;
* Treatment with any immunosuppressive therapy other than corticosteroids within 30 days prior to Screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-08 (Estimated)

PRIMARY OUTCOMES:
Serum levels of cytokines, troponin-T and D-dimer | Day 0, Day 2, Day 5, Day 10
  The endpoints are the change in the serum levels of cytokines, troponin-T and D-dimer from Day 0 to Day 5 of hospitalization, and from Day 0 to Day 10, as well as the area under the curve considering all measurements from Day 0 to Day 10.

SECONDARY OUTCOMES:
Time to clinical deterioration | Day 0 to Day 10
  Defined as time from randomization to mortality or worsening of the World Health Organization (WHO) Clinical Progression Scale, assessed by the increase of two points in this scale.
Adverse events | Day 0 to Day 10
  Cumulative incidence of adverse events
Severe adverse events | Day 0 to Day 10
  Cumulative incidence of severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, MD.PHD, Principal Investigator — State University of Campinas, Campinas, Brazil
Locations (2):
- Brazil (2):
  - Unicamp Clinical Hospital, Campinas, São Paulo
  - Hospital Estadual Sumaré, Sumaré, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tay MZ, Poh CM, Renia L, MacAry PA, Ng LFP. The trinity of COVID-19: immunity, inflammation and intervention. Nat Rev Immunol. 2020 Jun;20(6):363-374. doi: 10.1038/s41577-020-0311-8. Epub 2020 Apr 28. PMID 32346093
- [Result] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Result] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Result] Salama C, Han J, Yau L, Reiss WG, Kramer B, Neidhart JD, Criner GJ, Kaplan-Lewis E, Baden R, Pandit L, Cameron ML, Garcia-Diaz J, Chavez V, Mekebeb-Reuter M, Lima de Menezes F, Shah R, Gonzalez-Lara MF, Assman B, Freedman J, Mohan SV. Tocilizumab in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jan 7;384(1):20-30. doi: 10.1056/NEJMoa2030340. Epub 2020 Dec 17. PMID 33332779
- [Result] de Oliveira PG, Termini L, Durigon EL, Lepique AP, Sposito AC, Boccardo E. Diacerein: A potential multi-target therapeutic drug for COVID-19. Med Hypotheses. 2020 Nov;144:109920. doi: 10.1016/j.mehy.2020.109920. Epub 2020 Jun 1. PMID 32534337
- [Result] Martel-Pelletier J, Pelletier JP. Effects of diacerein at the molecular level in the osteoarthritis disease process. Ther Adv Musculoskelet Dis. 2010 Apr;2(2):95-104. doi: 10.1177/1759720X09359104. PMID 22870441
- [Result] Yang L, Li J, Xu L, Lin S, Xiang Y, Dai X, Liang G, Huang X, Zhu J, Zhao C. Rhein shows potent efficacy against non-small-cell lung cancer through inhibiting the STAT3 pathway. Cancer Manag Res. 2019 Feb 1;11:1167-1176. doi: 10.2147/CMAR.S171517. eCollection 2019. PMID 30774444
- [Result] Yang Y, Peng F, Wang R, Yange M, Guan K, Jiang T, Xu G, Sun J, Chang C. The deadly coronaviruses: The 2003 SARS pandemic and the 2020 novel coronavirus epidemic in China. J Autoimmun. 2020 May;109:102434. doi: 10.1016/j.jaut.2020.102434. Epub 2020 Mar 3. PMID 32143990
- [Result] Ragab D, Salah Eldin H, Taeimah M, Khattab R, Salem R. The COVID-19 Cytokine Storm; What We Know So Far. Front Immunol. 2020 Jun 16;11:1446. doi: 10.3389/fimmu.2020.01446. eCollection 2020. PMID 32612617
- [Result] Singh A, Strobbe D, Campanella M. Pyroptosis targeting via mitochondria: An educated guess to innovate COVID-19 therapies. Br J Pharmacol. 2022 May;179(10):2081-2085. doi: 10.1111/bph.15670. Epub 2021 Oct 10. PMID 34632567
- [Result] Ferreira AC, Soares VC, de Azevedo-Quintanilha IG, Dias SDSG, Fintelman-Rodrigues N, Sacramento CQ, Mattos M, de Freitas CS, Temerozo JR, Teixeira L, Damaceno Hottz E, Barreto EA, Pao CRR, Palhinha L, Miranda M, Bou-Habib DC, Bozza FA, Bozza PT, Souza TML. SARS-CoV-2 engages inflammasome and pyroptosis in human primary monocytes. Cell Death Discov. 2021 Mar 1;7(1):43. doi: 10.1038/s41420-021-00428-w. PMID 33649297
- [Result] Rodrigues TS, de Sa KSG, Ishimoto AY, Becerra A, Oliveira S, Almeida L, Goncalves AV, Perucello DB, Andrade WA, Castro R, Veras FP, Toller-Kawahisa JE, Nascimento DC, de Lima MHF, Silva CMS, Caetite DB, Martins RB, Castro IA, Pontelli MC, de Barros FC, do Amaral NB, Giannini MC, Bonjorno LP, Lopes MIF, Santana RC, Vilar FC, Auxiliadora-Martins M, Luppino-Assad R, de Almeida SCL, de Oliveira FR, Batah SS, Siyuan L, Benatti MN, Cunha TM, Alves-Filho JC, Cunha FQ, Cunha LD, Frantz FG, Kohlsdorf T, Fabro AT, Arruda E, de Oliveira RDR, Louzada-Junior P, Zamboni DS. Inflammasomes are activated in response to SARS-CoV-2 infection and are associated with COVID-19 severity in patients. J Exp Med. 2021 Mar 1;218(3):e20201707. doi: 10.1084/jem.20201707. PMID 33231615
- [Result] Vora SM, Lieberman J, Wu H. Inflammasome activation at the crux of severe COVID-19. Nat Rev Immunol. 2021 Nov;21(11):694-703. doi: 10.1038/s41577-021-00588-x. Epub 2021 Aug 9. PMID 34373622
- [Result] Fidelix TS, Macedo CR, Maxwell LJ, Fernandes Moca Trevisani V. Diacerein for osteoarthritis. Cochrane Database Syst Rev. 2014 Feb 10;2014(2):CD005117. doi: 10.1002/14651858.CD005117.pub3. PMID 24515444
- [Result] Huang M, Zong S-l and Zhang Q-y. The effect of food intake on the pk of rhein released from diacerein. Brazilian Journal of Pharmaceutical Sciences. 2020;56.
- [Result] Honvo G, Reginster JY, Rabenda V, Geerinck A, Mkinsi O, Charles A, Rizzoli R, Cooper C, Avouac B, Bruyere O. Safety of Symptomatic Slow-Acting Drugs for Osteoarthritis: Outcomes of a Systematic Review and Meta-Analysis. Drugs Aging. 2019 Apr;36(Suppl 1):65-99. doi: 10.1007/s40266-019-00662-z. PMID 31073924